CLINICAL TRIAL: NCT02932683
Title: Mednav: A Randomised Control Trial of Novice Users of Mednav a Neonatal Resuscitation Device at 0 and 7 Weeks Follow up.
Brief Title: MedNav: Improving Neonatal Life Support (NLS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: ChelseaNHS
Record Dates: First submitted 2016-10-12; First posted 2016-10-13 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Infant Showing No Response to Resuscitation
Keywords: Resuscitation; Neonatal; Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MedNav assisted resuscitators (Experimental): MedNav will be used to perform neonatal resuscitation on a mannequin and assessed after teaching and 7 weeks after intervention, following this a small group will be used as a cross over study.
  Interventions: Device: MedNav
- No MedNav resuscitators (No Intervention): Neonatal resuscitation will be performed on a mannequin (without the use of MedNav) and assessed after teaching and 7 weeks after intervention.

INTERVENTIONS:
Device: MedNav — MedNav is a tablet based platform that uses auditory and visual cues to prompt people to perform the correct steps in neonatal resuscitation.
  Arms: MedNav assisted resuscitators

SUMMARY:
This study was designed to evaluate if MedNav impacts the ability of novice resuscitators to perform Neonatal Life Support (NLS) in the simulated environment, and if this ability is maintained after a 7 week period. Testing the nul hypothesis that there is no difference in technical skill completion when performing neonatal resuscitation on a mannequin with or without MedNav, immediately after training or after a period of 7 weeks since the training episode.

DETAILED DESCRIPTION:
Novices resuscitators (Medical Students) were invited to attend a 2 hour teaching session on neonatal resuscitation.

To ensure that the differences in outcome of Neonatal Life Support (NLS) learning are attributable to MedNav only, a simple randomisation process was carried out just prior to testing, where candidates pulled out a folded piece of paper assigning them to either

1. No MedNav on performing NLS (control arm)
2. Assistance of MedNav when performing NLS

Blinding/masking was not possible for either the candidate or faculty as the testing process involved the use of a tablet device to display the MedNav system.

On entering the room, candidates stated whether they were using MedNav or not. Each candidate was given an identical neonatal resuscitation scenario and technical skills in neonatal resuscitation were assessed using a 12-point mark sheet adapted from the Neonatal Life Support course provided by the UK Resuscitation Council. After testing, all candidates were asked to assess their confidence in performing NLS using a seven point Likert scale.

Candidates were subsequently invited back for a follow-up session at 7 weeks. Testing of the same NLS scenario was undertaken with participants staying in their initial allocation groups. Again technical skills were assessed based on the UK resuscitation council mark sheet and candidates were asked to rate their confidence on NLS after.

For further analysis, a small sample of 9 students from the "non-MedNav" group were asked to perform NLS with the use of MedNav immediately after their secondary testing at 7 weeks. The investigators aim here was to assess if this crossover group had a significant improvement in their task completion owing largely to the use of MedNav.

ELIGIBILITY:
Inclusion Criteria:

Imperial Medical students Novice to Neonatal resuscitation Medical students with1 year of clinical experience.

Exclusion Criteria:

Previous Neonatal training,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-10; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Ability to perform Neonatal Resuscitation on a mannequin immediately and at 7 weeks following teaching. | 7 weeks
  Neonatal resuscitation will be assessed as defined by task completion based on an assessment sheet adapted from the resuscitation councils NLS course assessment.

SECONDARY OUTCOMES:
Confidence in performing neonatal resuscitation | 0 weeks and 7 weeks post teaching
  Confidence as marked on a 7 point Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Shane P Duffy, MBChB, Study Director — Chelsea and Westminster Hospital
Locations (1):
- Chelsea and Westminster NHS Foundation trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No